CLINICAL TRIAL: NCT04066088
Title: Dose Clinical Trial of Guanfacine Extended Release for the Reduction of Aggression and Self-injuries Behavior Associated With Prader-Willi Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI departure from institution
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19-00936
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Sham Comparator)
  Interventions: Other: Placebo
- GXR (Experimental): Immediately following the 8-week blinded randomized trial, an 8-week open-label continuation phase will be pursued to further define efficacy and tolerability of GXR, and to establish its safety with specific focus on metabolic profile.
  Interventions: Drug: Guanfacine extended release (GXR)

INTERVENTIONS:
Other: Placebo — Placebo will be administered same times as GXR
  Arms: Placebo
Drug: Guanfacine extended release (GXR) — The starting dose for all subjects will be 1 mg per day. If the medication is well-tolerated, the dose can be raised to 2 mg until day 28 and increased to 3mg for the remaining 4 weeks in the trial. The dose schedule will not be fixed; the treating clinician can delay a planned increase or lower the dose to manage adverse effects. At week 8, the study will be unblinded and subjects will continue treatment for 8 more weeks.
  Arms: GXR

SUMMARY:
This is a placebo-controlled clinical trial to assess the utility of Guanfacine Extended Release (GXR) in the management of patients with Prader Willi Syndrome (PWS) who have significant aggression or self-injury. The purpose of this trial is to establish the safety of GXR with a specific focus on metabolic effects.

DETAILED DESCRIPTION:
Prader-Willi syndrome is a genetic disorder due to loss of function of specific genes. In newborns, symptoms include weak muscles, poor feeding, and slow development. Beginning in childhood, the person becomes constantly hungry, which often leads to obesity and type 2 diabetes. Also, mild to moderate learning disability and behavioral problems are typical.

Guanfacine Extended Release (GXR), the investigational drug in this study would be the first study to evaluate the drug in patients with Prader Willi Syndrome. "Investigational" means it is not approved by the Food and Drug Administration (FDA) to treat Prader Willi Syndrome. However, Guanfacine Extended Released (GXR) is an FDA approved drug used to treat children and adolescents with hypertension and attention deficit hyperactivity disorder (ADHD). GXR is thought to respond to parts of the brain that lead to strengthening working memory, reducing distraction, improving attention and impulse control. GXR is generally considered safe for children as long as it is used according to the dosing instructions (up to 4mg) of a qualified medical professional.

ELIGIBILITY:
Inclusion Criteria:

* 6 and 35 years of age
* diagnosis of PWS confirmed by genetic testing.
* rating of moderate or above on the Clinical Global Impression- Severity Scale will be required for entry.

Exclusion Criteria:

* Subjects with a positive pregnancy test, swallowing difficulty, and/or presenting with active psychosis or mania will be excluded.
* Individuals with pre-existing, clinically significant bradycardia (< 8 years: <64 bpm; 8 to 12 years: <59 bpm; 12 to 16 years: <53 bpm) or hypotension, defined as 5th percentile for height and gender,26 will be excluded from the study.
* Subjects receiving antipsychotic medications due to a documented history of psychosis or bipolar disorder will be allowed to continue taking the medication without dosage modification.
* Growth hormone, thyroid hormone replacement treatment, and non-psychiatric medicines will be allowed to continue.
* N-Acetyl Cysteine and anticonvulsant medication (only if prescribed for seizures) will be allowed to continue, with specific instructions to not make any dosage changes during the clinical trial.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
CGI-I scale rating | 19 Weeks
  A positive clinical response will be determined by a rating of 1 or 2 (Very much/Much improved) on the CGI-I scale at the end of the blinded trial.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist | 19 Weeks
  Consists of 2 subscales; irritability (15 items) and hyperactivity/noncompliance (16 items).
Self-Injury Trauma scale | 19 Weeks
  SHI scores of 5 or greater were found to be indicative of borderline personality disorder. Part 1 is ranking based on the number of wounds 1=one would (common in a mild SIB but rare in a severe case) 2=two or four wounds (common) and 3=five or more wounds (rare). Injury severity is scored on a subjective basis with labels such as "mild" "moderate" and "severe" accompanied by descriptions of the observed state of the anatomy. Part 3 is the Estimate of Current Risk.
Modified Overt Aggression Scale | 19 Weeks
  four-part behavior rating scale used to evaluate and document the "frequency and severity" of aggressive episodes.[1] The rating scale is made up of four categories; verbal aggression, aggression against objects, aggression against self, and aggression against others

CONTACTS AND LOCATIONS:
Overall Officials: Deepan Singh, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States